CLINICAL TRIAL: NCT03383081
Title: A Clinical Research on the Safety/Efficacy of Human Umbilical Cord Mesenchymal Stem Cells（19#iSCLife®-OA） Therapy for Patients With Osteoarthritis
Brief Title: The Safety/Efficacy of hUC Mesenchymal Stem Cells（19#iSCLife®-OA） Therapy for Patients With Osteoarthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sclnow Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCLnow-XY-02
Record Dates: First submitted 2017-12-12; First posted 2017-12-26 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis, mesenchymal stem cell
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Injections, Intra-Articular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose mesenchymal stem cells (Experimental): Low dose group: intra-articular injection with human umbilical cord mesenchymal stem cells (SCLnow 19#)
  Interventions: Biological: Low dose mesenchymal stem cells; Procedure: Intraarticular injection
- High dose mesenchymal stem cells (Experimental): High dose group: intra-articular injection with human umbilical cord mesenchymal stem cells (SCLnow 19#)
  Interventions: Biological: High dose mesenchymal stem cells; Procedure: Intraarticular injection
- Control groups (No Intervention): No intervention

INTERVENTIONS:
Biological: Low dose mesenchymal stem cells — Human umbilical cord mesenchymal stem cells (SCLnow 19#): group A, 1 * 10^7 cells (5ml);
  Arms: Low dose mesenchymal stem cells
Biological: High dose mesenchymal stem cells — Human umbilical cord mesenchymal stem cells (SCLnow 19#): group B, 2 * 10^7 cells (5ml)
  Arms: High dose mesenchymal stem cells
Procedure: Intraarticular injection — Intraarticular injection with human umbilical cord mesenchymal stem cells (SCLnow 19#) with different dose group
  Arms: High dose mesenchymal stem cells; Low dose mesenchymal stem cells

SUMMARY:
The purpose of this study is verify the efficacy and safety of Human Umbilical Cord Mesenchymal Stem Cells (UC-MSC) therapy for patients with Osteoarthritis, and in addition, provide basis for exploring the treatment regimen of UC-MSC therapy in different degree of cartilage defect disease

DETAILED DESCRIPTION:
This is a random, open label, and parallel controled experiment. All patients are selected and sign consent forms, then divided into 3 groups. Doctors collect the basic information of patient. All patients receive laboratory and image examination as baseline. Then, they will give cell treatment based on the clinical protocol. Doctors have follow-up visit on 2 weeks, 1, 2, 3, 6, and 12 months after treatment, and do safety and efficacy evaluation.

Safety evaluation. Researcher collect all examination data of patients and compare with each groups. The safety tests including blood routine, urine routine, hepatorenal function, C reactive protein, erythrocyte sedimentation rate, and tumor marker, etc.

Efficacy evaluation. Based on Lysholm, the international knee documentation committee (IKDC) knee evaluation form, and Visual Analogue Scale/Score (VAS) to examine the change/improvement of knee joint function. By Magnetic Resonance Imaging (MRI) examination, grade patients with Kellgren-Lawrence Grading Scale, Assessment of Preoperative Cartilage Defect Severity (AMADEUS), and observe the change/improvement of patient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Knee Osteoarthritis by Kellgren and Lawrence Grading Scale, classified with Grade 2-3
* Confirm with cartilage injury,articular cartilage part or full-thickness injury, by MR (Magnetic Resonance)
* Age <70, no serious organ dysfunction
* Over 2 years knee pain or no very effective with conservative treatments
* Knee pain of VAS (visual analog scale score) is 4 or higher
* Normal hepatic and renal function, no history of gout, rheumatoid arthritis, and autoimmune diseases, etc.
* Understand and sign the consent form of this study

Exclusion Criteria:

* Refuse to sign the consent form, or cannot keep follow-up visit
* Age >70; Age <70, but with multiple organ failure
* Unstable vital signs (breath, blood pressure, pulse)
* Combined with knee ligament (anterior and the posterior cruciate ligament, medial and lateral collateral ligament) rupture, laxity, etc.
* Serious bleeding tendency, poor coagulation function (PTA <35%)
* Pregnant or breast feeding women, or positive pregnancy test in 7 days before treatment
* Participate other clinical experiments in 3 months
* With progressing malignant tumor
* Combined with shock and critically ill patients
* With mental disease, cannot
* With history of knee joint infection, surgery, and radiotherapy
* With immunosuppressive agents treatment in 6 weeks
* Injection with hormones and sodium hyaluronate in joint in 3 months
* Overweight expressed as body mass index (BMI) >35
* With skin disease around knee joint
* With Immunodeficiency disease, including long term use immunosuppressive agents patients
* Combined with serious infection
* With some other conditions that doctor propose not to participate

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Kellgren-Lawrence Grading Scale | 12 months
  Using Magnetic Resonance Imaging (MRI) examination, and based on the images of bilateral knee joint, grade by Kellgren-Lawrence Grading Scale. Kellgren-Lawrence Grading Scale is a method of classifying the severity of knee osteoarthritis (OA).
  Grade 0: No radiographic features of osteoarthritis; Grade 1: Possible joint space narrowing (normal joint space is at least 2 mm at the superior acetabulum) and osteophyte formation; Grade 2: Definite osteophyte formation with possible joint space narrowing; Grade 3: Multiple osteophytes, definite joint space narrowing, sclerosis and possible bony deformity; Grade 4: Large osteophytes, marked joint space narrowing, severe sclerosis and definite bony deformity.

SECONDARY OUTCOMES:
Assessment of Preoperative Cartilage Defect Severity (AMADEUS) | 12 months
  Using Magnetic Resonance Imaging (MRI) examination to diagnose patients by Assessment of Preoperative Cartilage Defect Severity (AMADEUS).
Lysholm scoring | 12 months
  Using Lysholm Knee Scoring Scale to grade the knee function of patients, and examine the changes or improvement compare to baseline.
The international knee documentation committee (IKDC) knee evaluation form | 12 months
  The international knee documentation committee knee evaluation form is used to assess the knee function of patients, examine the changes or improvement compare to baseline.
Visual Analogue Scale/Score（VAS） | 12 months
  Using Visual Analogue Scale/Score for pain to examine the change/improvement of knee joint function.

CONTACTS AND LOCATIONS:
Overall Officials: Hongbin Lu, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China